CLINICAL TRIAL: NCT02243579
Title: A Phase 2 Study of MK-3475 for the Treatment of Relapsed/Refractory Mycosis Fungoides/Sezary Syndrome
Brief Title: Pembrolizumab in Treating Patients With Relapsed or Refractory Stage IB-IVB Mycosis Fungoides or Sezary Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2014-00709; NCI-2014-00709 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CITN-10 (Other: Cancer Immunotherapy Trials Network); CITN-10 (Other: CTEP); P30CA015704 (NIH); U01CA154967 (NIH)
Record Dates: First submitted 2014-09-16; First posted 2014-09-18 (Estimated); Results first posted 2019-02-05 (Actual); Last update posted 2019-09-20 (Actual); Status verified 2019-08

CONDITIONS: Recurrent Mycosis Fungoides and Sezary Syndrome; Refractory Mycosis Fungoides and Sezary Syndrome; Stage IB Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IIA Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IIB Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IIIA Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IIIB Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IVA Mycosis Fungoides and Sezary Syndrome AJCC v7; Stage IVB Mycosis Fungoides and Sezary Syndrome AJCC v7
MeSH Terms: conditions — Mycosis Fungoides; Sezary Syndrome | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Treatment (pembrolizumab) (Experimental): Patients receive pembrolizumab IV over 30 minutes on day 1. Courses repeat every 3 weeks for up to 2 years (6 months for patients achieving CR) in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Biological: Pembrolizumab

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Biological: Pembrolizumab — Given IV
  Other Names: Keytruda; Lambrolizumab; MK-3475; SCH 900475

SUMMARY:
This phase II trial studies how well pembrolizumab works in treating patients with stage IB-IVB mycosis fungoides or Sezary syndrome that has returned after a period of improvement or has not responded to at least one type of treatment. Monoclonal antibodies, such as pembrolizumab, may block cancer growth in different ways by targeting certain cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the response rate of MK-3475 (pembrolizumab) in subjects with relapsed/refractory mycosis fungoides/Sezary syndrome (MF/SS).

SECONDARY OBJECTIVES:

I. To explore the clinical activity of MK-3475 in subjects with relapsed/refractory MF and SS with respect to the following endpoints: duration of response (DOR); progression-free survival (PFS); overall survival (OS).

OUTLINE:

Patients receive pembrolizumab intravenously (IV) over 30 minutes on day 1. Courses repeat every 3 weeks for up to 2 years (6 months for patients achieving complete response [CR]) in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 30 days and then every 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* This trial will include subjects with stage IB-IVB MF/SS (maximal stage since diagnosis will determine eligibility), and who have relapsed, are refractory, or progressed after at least one standard systemic therapy; current disease stage at time of entry will also be documented but will not be used for eligibility
* Subjects must have the following minimum wash-out and adverse event (AE) recovery period from previous treatments without treatment between documentation of relapse/progression and enrollment of specifically:

  * >= 2 weeks for local radiation therapy
  * >= 4 weeks for systemic cytotoxic anticancer agents, anticancer investigational agents that are not defined as immunotherapy, or for tumor-targeting monoclonal antibodies (mAbs) with the exception of alemtuzumab for which the washout is at least 8 weeks
  * >= 15 weeks for anti-cluster of differentiation (CD)137 or anti-cytotoxic T-lymphocyte-associated protein 4 (CTLA-4) (including ipilimumab or any other antibody or drug specifically targeting T-cell co-stimulation or checkpoint pathways)
  * >= 2 weeks from resolution (i.e., =< grade 1 or at baseline) from AEs due to procedures performed or therapeutic agents administered
  * >= 2 weeks for retinoids, interferons, vorinostat, romidepsin, denileukin diftitox, and therapeutic doses of oral corticosteroids (physiologic replacement doses of oral corticosteroids are allowed, topical corticosteroids are allowed)
  * >= 2 weeks for phototherapy
  * >= 1 week for topical therapy (including retinoid, nitrogen mustard, or imiquimod)
* Have a performance status of 0 or 1 on the Eastern Cooperative Oncology Group (ECOG) performance scale
* Life expectancy of at least 6 months
* Performed within 10 days of treatment initiation: Leukocytes >= 2,000/mcL
* Performed within 10 days of treatment initiation: Absolute neutrophil count >= 1,500/mcL
* Performed within 10 days of treatment initiation: Platelets >= 100,000/mcL
* Performed within 10 days of treatment initiation: Hemoglobin >= 9 g/dL OR >= 5.6 mmol/L
* Performed within 10 days of treatment initiation: Serum total bilirubin =< 1.5 x upper limit of normal (ULN) OR direct bilirubin =< ULN for subjects with total bilirubin levels > 1.5 ULN
* Performed within 10 days of treatment initiation: Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT]) and alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 2.5 x ULN OR =< 5 x ULN for patients with liver metastases
* Performed within 10 days of treatment initiation: Serum creatinine =< 1.5 x ULN OR measured or calculated creatinine clearance >= 60 mL/min for subject with creatinine clearance (CrCl) levels > 1.5 x institutional ULN (glomerular filtration rate [GFR] can also be used in place of creatinine or CrCl)
* Performed within 10 days of treatment initiation: International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy in which case the INR or PT must be within the therapeutic range of intended use for the anticoagulant
* Performed within 10 days of treatment initiation: Activated partial thromboplastin time (aPTT) =< 1.5 x ULN unless subject is receiving anticoagulant therapy in which case the aPTT must be within the therapeutic range of intended use for the anticoagulant
* Performed within 10 days of treatment initiation: Thyroid stimulating hormone (TSH) within institutional limits (ie: normal); if TSH is greater or less than institutional limits patients may participate if their thyroxine (T4) is within normal limits (WNL); patients may be on a stable dose of replacement thyroid medication; dose adjustments are allowed if needed
* Patients must provide tissue from a punch biopsy of the skin at baseline, at the time of a clinical event (at the time of response, progression or appearance of a new lesion) and at the end of treatment; additional punch biopsies every 3 cycles are optional; an archival tissue sample is optional
* Have measurable disease based on modified severity-weighted assessment tool (mSWAT); tumor lesions situated in a previously irradiated area are considered measurable if progression has been demonstrated in such lesions
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) from the time of the pre-study visit, through the course of the study and for 120 days after the last dose of study medication

  * Female patients of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of study medication; if the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required
  * Female patients of childbearing potential should be willing to use 2 methods of birth control or be surgically sterile, or abstain from heterosexual activity from the time of the pre-study visit, through the course of the study and for 120 days after the last dose of study medication; patients of childbearing potential are those who have not been surgically sterilized or have not been free from menses for > 1 year
  * Should a woman become pregnant or suspect she is pregnant while she is participating in this study, she should inform her treating physician immediately; men treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and 4 months after completion of MK-3475 administration
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or targeted small molecule therapy within 4 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 4 weeks earlier

  * Note: patients with =< grade 2 neuropathy are an exception to this criterion and may qualify for the study
  * Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy
* Patients who are currently participating in or have participated in a study of an investigational agent or using an investigational device within 4 weeks of the first dose of treatment
* Has a diagnosis of immunodeficiency or is receiving therapeutic systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of trial treatment
* Has had a prior monoclonal antibody within 4 weeks prior to study day 1 or who has not recovered (i.e., =< grade 1 or at baseline) from AEs due to agents administered more than 4 weeks earlier
* Has a known additional malignancy that is progressing or requires active treatment; exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy
* Patients with known brain metastases should be excluded from this clinical trial

  * Patients with carcinomatous meningitis should also be excluded
  * Patients with previously treated brain metastases may participate provided they are stable (without evidence of progression by imaging for at least 4 weeks prior to the first dose of trial treatment and any neurologic symptoms have returned to baseline), have no evidence of new or enlarging brain metastases, and are not using steroids for at least 7 days prior to trial treatment
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to MK-3475
* Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents; patients with vitiligo or resolved childhood asthma/atopy would be an exception to this rule; patients that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study; the use of physiologic doses of corticosteroids may be approved after consultation with the protocol principal investigator (PI) and Cancer Immunotherapy Trials Network (CITN); patients with hypothyroidism stable on hormone replacement or Sjogren's syndrome will not be excluded from the study
* Has a history or current evidence of any condition, therapy, or laboratory abnormality that might confound the results of the trial, interfere with the patient's participation for the full duration of the trial, or is not in the best interest of the patient to participate, in the opinion of the treating investigator
* Has known psychiatric or substance abuse disorders that would interfere with cooperation with the requirements of the trial
* Has received prior therapy with an anti-programmed cell death (PD)-1, anti-PD-ligand (L)1, anti-PD-L2
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, interstitial lung disease or active, non-infectious pneumonitis, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* History of other pulmonary disease such as emphysema or chronic obstructive pulmonary disease, (forced expiratory volume in one second [FEV1] < 60% of predicted for height and age); pulmonary function tests (PFTs) are required in patients with prolonged smoking history or symptoms of respiratory dysfunction
* Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the pre-study visit through 120 days after the last dose of trial treatment; breastfeeding should be discontinued if the mother is treated with MK-3475

  * Men and non-pregnant, non-breast-feeding women may be enrolled if they are willing to use 2 methods of birth control or are considered highly unlikely to conceive; highly unlikely to conceive is defined as 1) surgically sterilized, or 2) postmenopausal (a woman who is >= 45 years of age and has not had menses for greater than 1 year will be considered postmenopausal), or 3) not heterosexually active for the duration of the study; the two birth control methods can be barrier method or a barrier method plus a hormonal method to prevent pregnancy; patients should start using birth control from the time of the pre-study visit, through the course of the study and for 120 days after the last dose of study medication; the following are considered adequate barrier methods of contraception: diaphragm, condom (by the partner), copper intrauterine device, sponge, or spermicide; appropriate hormonal contraceptives will include any registered and marketed contraceptive agent that contains an estrogen and/or a progestational agent (including oral, subcutaneous, intrauterine, or intramuscular agents)
  * Patients should be informed that taking the study medication may involve unknown risks to the fetus (unborn baby) if pregnancy were to occur during the study; in order to participate in the study they must adhere to the contraception requirement (described above) for the duration of the study and during the follow-up period; if there is any question that a patient will not reliably comply with the requirements for contraception, that patient should not be entered into the study
  * If a patient inadvertently becomes pregnant while on treatment with MK-3475, the patient will immediately be removed from the study; the site will contact the patient at least monthly and document the patient's status until the pregnancy has been completed or terminated; the outcome of the pregnancy will be reported without delay and within 24 hours if the outcome is a serious adverse experience (e.g., death, abortion, congenital anomaly, or other disabling or life-threatening complication to the mother or newborn); the study investigator will make every effort to obtain permission to follow the outcome of the pregnancy and report the condition of the fetus or newborn; if a male patient impregnates his female partner the study personnel at the site must be informed immediately and the pregnancy reported and followed
* Patients who are human immunodeficiency virus (HIV) positive may participate IF they meet the following eligibility requirements:

  * They must be stable on their anti-retroviral regimen, and they must be healthy from an HIV perspective
  * They must have a CD4 count of greater than 250 cells/mcL
  * They must not be receiving prophylactic therapy for an opportunistic infection
* Has known active hepatitis B (e.g., hepatitis B surface antigen [HBsAg] reactive) or hepatitis C (e.g., hepatitis C virus [HCV] ribonucleic acid [RNA] [qualitative] is detected)
* Has received a live vaccine within 30 days prior to the first dose of trial treatment
* Has a known human T-lymphotropic virus type 1 (HTLV) infection
* Patient has a history of (non-infectious) pneumonitis that required steroids or current pneumonitis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-10-15 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Youn Kim, Principal Investigator — Cancer Immunotherapy Trials Network
Locations (8):
- United States (8):
  - Stanford Cancer Institute Palo Alto, Palo Alto, California
  - Yale University, New Haven, Connecticut
  - Moffitt Cancer Center, Tampa, Florida
  - Johns Hopkins University/Sidney Kimmel Cancer Center, Baltimore, Maryland
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Ohio State University Comprehensive Cancer Center, Columbus, Ohio
  - University of Pennsylvania/Abramson Cancer Center, Philadelphia, Pennsylvania
  - Seattle Cancer Care Alliance, Seattle, Washington

REFERENCES:
- [Derived] Phillips D, Matusiak M, Gutierrez BR, Bhate SS, Barlow GL, Jiang S, Demeter J, Smythe KS, Pierce RH, Fling SP, Ramchurren N, Cheever MA, Goltsev Y, West RB, Khodadoust MS, Kim YH, Schurch CM, Nolan GP. Immune cell topography predicts response to PD-1 blockade in cutaneous T cell lymphoma. Nat Commun. 2021 Nov 18;12(1):6726. doi: 10.1038/s41467-021-26974-6. PMID 34795254
- [Derived] Khodadoust MS, Rook AH, Porcu P, Foss F, Moskowitz AJ, Shustov A, Shanbhag S, Sokol L, Fling SP, Ramchurren N, Pierce R, Davis A, Shine R, Li S, Fong S, Kim J, Yang Y, Blumenschein WM, Yearley JH, Das B, Patidar R, Datta V, Cantu E, McCutcheon JN, Karlovich C, Williams PM, Subrahmanyam PB, Maecker HT, Horwitz SM, Sharon E, Kohrt HE, Cheever MA, Kim YH. Pembrolizumab in Relapsed and Refractory Mycosis Fungoides and Sezary Syndrome: A Multicenter Phase II Study. J Clin Oncol. 2020 Jan 1;38(1):20-28. doi: 10.1200/JCO.19.01056. Epub 2019 Sep 18. PMID 31532724

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pembrolizumab)
Started | 24
Completed | 4
Not Completed | 20

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 15
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 20
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate (ORR), Defined as a Confirmed Partial Response (PR) or Complete Response (CR) Using Global Assessment Standard Response Criteria for Mycosis Fungoides and Sezary Syndrome
Description: A generalized linear model for the objective response rate used a binominal error distribution. The model included as covariates all available baseline predictors of the missing outcomes.
Time Frame: Up to 3.2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 24
Participants
  Confirmed Complete Response | 2
  Confirmed Partial Response | 7
  Stable Disease | 9
  Progressive Disease | 6

2. Secondary Outcome: Duration of Response
Description: Was estimated using the Kaplan-Meier method (Duration of Response Probability).
Time Frame: The time interval between the date of first response (CR/PR) and the date of progression as assessed by standard Mycosis Fungoides and Sezary Syndrome response criteria, assessed at 26 and 52 weeks
Measure: Number; unit: Duration of Response Probability
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 9
Duration of Response Probability
  26 weeks | 1.0
  52 weeks | 0.8571

3. Secondary Outcome: Progression Free Survival (PFS)
Description: Was estimated using the Kaplan-Meier method (Progression Free Survival Probability).
Time Frame: The time from allocation to the first documented disease progression or death due to any cause, whichever occurs first, assessed at 26 and 52 weeks
Measure: Number; unit: Progression Free Survival Probability
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 24
Progression Free Survival Probability
  26 weeks | 0.7380
  52 weeks | 0.6457

4. Secondary Outcome: Overall Survival (OS)
Description: Was estimated using the Kaplan-Meier method (Overall Survival Probability).
Time Frame: The time from randomization to death due to any cause, assessed at 52, 104 and 156 weeks
Measure: Number; unit: Overall Survival Probability
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 24
Overall Survival Probability
  52 weeks | 0.95
  104 weeks | 0.7917
  156 weeks | 0.5429

5. Secondary Outcome: Time to Onset of First Drug-related Toxicity
Description: Summary statistics (mean and SD) for time to onset of first drug-related toxicity was provided.
Time Frame: Up to 4 years
Population: Patients with drug-related toxicities included in the analysis
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 22
Days | 64.5 (121.3)

6. Secondary Outcome: Incidence of Adverse Events Graded Using the Common Terminology Criteria for Adverse Events Version 5.0
Description: Adverse events were summarized as counts and frequencies by toxicity grade.
Time Frame: Up to 4 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (Pembrolizumab)
Number analyzed (Participants) | 24
Participants
  Maximum Toxicity Grade 1 | 2
  Maximum Toxicity Grade 2 | 7
  Maximum Toxicity Grade 3 | 9
  Maximum Toxicity Grade 4 | 6

ADVERSE EVENTS:
Time Frame: Up to 4 years
Arm/Group | Treatment (Pembrolizumab)
All-Cause Mortality (participants affected / at risk) | 7/24
Serious Adverse Events (participants affected / at risk) | 11/24
Other Adverse Events (participants affected / at risk) | 24/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=24)
Atrial Fibrillation (Cardiac disorders) | 1
Heart Failure (Cardiac disorders) | 1
Corneal Ulcer (Eye disorders) | 1
Periorbital Edema (Eye disorders) | 1
Colitis (Gastrointestinal disorders) | 1
Colonic obstruction (Gastrointestinal disorders) | 1
Duodenitis (Gastrointestinal disorders) | 1
Edema face (General disorders) | 1
Fatigue (General disorders) | 1
Anaphylaxis (Immune system disorders) | 1
Lung Infection (Infections and infestations) | 1
Sepsis (Infections and infestations) | 1
Urinary Tract Infection (Infections and infestations) | 2
Alanine Aminotransferase increased (Investigations) | 1
Aspartate Aminotransferase increased (Investigations) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Confusion (Psychiatric disorders) | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pneuminitis (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary Edema (Respiratory, thoracic and mediastinal disorders) | 1
Hypertension (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Pembrolizumab) (N=24)
Anemia (Blood and lymphatic system disorders) | 7
Low Hemoglobin (Blood and lymphatic system disorders) | 1
Vertigo (Ear and labyrinth disorders) | 2
Blurred Vision (Eye disorders) | 1
Keratitis (Eye disorders) | 1
Abdominal Pain (Gastrointestinal disorders) | 1
Colonic hemorrhage (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhea (Gastrointestinal disorders) | 3
Nausia (Gastrointestinal disorders) | 2
Vomiting (Gastrointestinal disorders) | 1
Chills (General disorders) | 1
Edema face (General disorders) | 2
Edema limbs (General disorders) | 4
Edema trunk (General disorders) | 1
Fatigue (General disorders) | 7
Fever (General disorders) | 2
Weakness (General disorders) | 1
Weakness (grade decrease) (General disorders) | 1
Firm tender lump on his left lateral thigh, no trauma to the area (General disorders) | 1
Generalized edema (General disorders) | 1
Malaise (General disorders) | 1
Pain (General disorders) | 1
Inflammation/Flare reaction (Immune system disorders) | 1
Conjunctivitis (Infections and infestations) | 1
Esophageal infection (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Infection S/P scheduled Mohs surgery (Infections and infestations) | 1
Right lower leg infection related to approved radiation and wound care (Infections and infestations) | 1
Mucosal infection (thrush) (Infections and infestations) | 1
Mucosal infection - thrush (Infections and infestations) | 1
Upper eyelid infection (Infections and infestations) | 1
otitis externa (Infections and infestations) | 1
rash pustular (Infections and infestations) | 1
Skin infection (Infections and infestations) | 2
Soft tissue infection (Infections and infestations) | 1
Upper respiratory infection (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Infusion related reaction (Injury, poisoning and procedural complications) | 2
Alanine aminotransferase increased (Investigations) | 2
Alkaline phosphatase inceased (Investigations) | 1
Aspartate aminotransferase increased (Investigations) | 2
Blood bilirubin increased (Investigations) | 2
Cardiac troponin T increased (Investigations) | 1
Creatinine increased (Investigations) | 4
Investigations (Investigations) | 1
Lymphocyte count decreased (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Weight gain (Investigations) | 1
Weight loss (Investigations) | 2
white blood cell decreased (Investigations) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 6
Hyperkalemia (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 5
Hypoalbuminemia (Metabolism and nutrition disorders) | 2
Hypocalcemia (Metabolism and nutrition disorders) | 5
Hypokalemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Muscle weakness lower limb (Musculoskeletal and connective tissue disorders) | 1
Herniated disc (Musculoskeletal and connective tissue disorders) | 1
neck pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3
BCC right leg (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
SCC forehead (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Ataxia (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Tremor (Nervous system disorders) | 1
Anxiety (Psychiatric disorders) | 1
Confusion (Psychiatric disorders) | 3
Insomnia (Psychiatric disorders) | 2
Nephrolithiasis (Renal and urinary disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Horseness (Reproductive system and breast disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Bilateral pulmonary infiltrates (Respiratory, thoracic and mediastinal disorders) | 1
Sinus inflammation (Respiratory, thoracic and mediastinal disorders) | 1
Alopecia (Skin and subcutaneous tissue disorders) | 3
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 3
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Skin eruption/flare, rash (Skin and subcutaneous tissue disorders) | 1
immune mediated flare reaction on the face (Skin and subcutaneous tissue disorders) | 1
pustular rash (Skin and subcutaneous tissue disorders) | 1
Mild skin peeling (Skin and subcutaneous tissue disorders) | 1
Erythroderma (Skin and subcutaneous tissue disorders) | 1
Night sweats (Skin and subcutaneous tissue disorders) | 1
Skin flare (Skin and subcutaneous tissue disorders) | 1
Excess skin peeling (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Scheduled Mohs surgery (Surgical and medical procedures) | 1
Hot flashes (Vascular disorders) | 1
Hypertension (Vascular disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-08): https://cdn.clinicaltrials.gov/large-docs/79/NCT02243579/Prot_SAP_000.pdf